CLINICAL TRIAL: NCT04285619
Title: Effectiveness of a Physiotherapy Intervention With Flossing Conditioned by the Verbal Suggestion of an Expectation About Ankle Functionality in Amateur Runners. A Randomized Clinical Trial.
Brief Title: Physiotherapy Intervention With Flossing Conditioned by Verbal Suggestion About Ankle Functionality in Amateur Runners
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLOSSINGRUN
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Running
Keywords: Amateur runners; Ankle dorsiflexion; Flossing; Expectancy; Randomized clinical trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 10 minutes and a weekly intervention will take place over 3 weeks. The intervention by flossing will be carried out following the application protocol described by the manufacturer for the application of flossing on the ankle. Before the intervention, participants will perform a standard warm-up: 10 minutes of exercise bike at a moderate intensity
  Interventions: Other: Positive expectation
- Control group (Active Comparator): Each session will last 10 minutes and a weekly intervention will take place over 3 weeks. The intervention by flossing will be carried out following the application protocol described by the manufacturer for the application of flossing on the ankle. Before the intervention, participants will perform a standard warm-up: 10 minutes of exercise bike at a moderate intensity
  Interventions: Other: Neutral expectation

INTERVENTIONS:
Other: Positive expectation — After heating, the physiotherapist will apply the bandage with flossing on both ankles, using 2 Voodoo Floss Bands (Power Guidance model). The distal to proximal bandage will begin with a tension of 50-70% and each lap of the bandage will cover 50% of the previous lap. There will be 3 figures of 8 that will cover the hindfoot and the distal third of the leg.
  With the bandage applied on both feet, the runners will perform plantar flexion and active dorsal flexion movements in a range of complete joint movement with both ankles, at a constant rate of 2 seconds of plantar flexion, followed by another 2 of dorsal flexion, during A period of 2 minutes. Next, the therapist will remove the bandages and the athlete will walk barefoot for a minute, to restore normal blood flow.
  During the first application of the bandage, the investigator will induce the positive expectation through a standardized phrase for all subjects
  Arms: Experimental group
Other: Neutral expectation — After heating, the physiotherapist will apply the bandage with flossing on both ankles, using 2 Voodoo Floss Bands (Power Guidance model). The distal to proximal bandage will begin with a tension of 50-70% and each lap of the bandage will cover 50% of the previous lap. There will be 3 figures of 8 that will cover the hindfoot and the distal third of the leg.
  With the bandage applied on both feet, the runners will perform plantar flexion and active dorsal flexion movements in a range of complete joint movement with both ankles, at a constant rate of 2 seconds of plantar flexion, followed by another 2 of dorsal flexion, during A period of 2 minutes. Next, the therapist will remove the bandages and the athlete will walk barefoot for a minute, to restore normal blood flow.
  During the first application of the bandage, the researcher will not induce any expectations to the athletes.
  Arms: Control group

SUMMARY:
Limited ankle functionality is one of the main causes of runner injuries. The use of flossing techniques are used to improve functionality. The administration of an expectation can modulate corticospinal excitability, improving the therapeutic response.

The objective of the study is to evaluate the effect of inducing a positive expectation along with the application of flossing on the ankle functionality in healthy amateur runners.

Randomized clinical study, single blind, with follow-up period. 20 runners will be randomized to the two study groups: experimental (flossing technique with a positive expectation) and control (flossing technique with a neutral expectation). The study variables will be: dorsal ankle flexion (Weigh Bearing Lunge Test), isometric force in plantar ankle flexion (dynamometry), elastic-explosive force (Countermovement Jump) and stability (Y Balance Test). Using a Shapiro-Wilks analysis, the sample distribution will be calculated. The changes after each evaluation will be analyzed with the t-student test of related samples and through an ANOVA of repeated measures the intra and intersubject effect will be observed. The effect size will be calculated using Cohen's formula.

It is expected to obtain changes in the variables between both groups and in the group / time interaction, which suggest an effect of the expectation on corticospinal excitability in healthy athletes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer amateur runners
* Both sexes
* Aged between 18 and 35 years
* That they practice a recreational career for a minimum of 2 days per week, with a duration of 60 minutes per session and an experience of 1 year in this sports field
* Obtain a score equal to or greater than 96 in the VISA-A questionnaire and at least 96% in the FAAM-Sp

Exclusion Criteria:

* Subjects who have suffered an injury to the lower limb in the last 6 months
* Have peripheral skin, vascular, muscle or nerve lesions, a history of cardiovascular or metabolic disease and coagulation problems at the time of the study
* That have been previously treated with flossing; who have taken antiinflammatory drugs in the last week
* Have not signed the informed consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline dorsal ankle flexion after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be assessed with the Weigh Bearing Lunge Test. The Dorsiflex iPhone application will be used. The subject will stand in stride position, with the dominant leg more advanced, to perform the measurement on it. Next, the evaluator will support the vertical and parallel iPhone on the tibia, so that the upper corner of the phone is in contact with the anterior tibial tuberosity and along the diaphysis. The investigator will give 5 seconds to achieve maximum dorsal ankle flexion, advancing the knee as far as possible without the heel detaching from the ground. Next, the same procedure will be performed on the contralateral member. This measurement will be performed 3 times, alternately on each ankle, with a 30-second wait interval, and the average of each ankle will be calculated to obtain the definitive value of the measurement (34). The unit of measure will be degrees with decimals.

SECONDARY OUTCOMES:
Change from baseline isometric force after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  This variable will be measured in Newtons (N), with a manual digital dynamometer (wireless microFET®2 model). The athlete will be placed supine with the knees extended and the ankles in plantar flexion relaxed. The dynamometer will be placed over the head of the metatarsals of the foot. The runner will be instructed to gradually increase his strength for 3 seconds and to make maximum force against the dynamometer for another 2 seconds only with his ankle withdrawing his foot quickly. The record will be repeated 3 times, with 30 seconds between repetitions, to avoid the effects of post-activation enhancement accrued from the realization of a maximum voluntary isometric force. The average of the 3 will be obtained to calculate the measurement value.
Change from baseline elastic-explosive force after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be calculated with the Countermovement Jump test. The result is measured with the jump height in centimeters (cm) or the flight time in seconds (sg). We will measure the height of the jump (cm) with the MyJump application for iPhone. The runner will stand in standing position with feet apart at the height of the hips, straight legs and hands resting on the hips. The evaluator will focus the feet to record. The participant will be asked to jump as high as possible, without separating the hands from the hips, keeping the legs straight during the flight and landing simultaneously with both feet. Recording will pause and wait 30 seconds to repeat the jump. There will be 3 jumps in total and the average of them will be made to determine the final value in cm.
Change from baseline stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The evaluation will be measured in centimeters using the Star Excursion Balance Test. This test consists of moving a moving part with the foot, in monopodal support, on 3 axes of movement, separated from each other 135º - 90º - 135º; anterior (0º), posteromedial (135º) and posterolateral (225º). The maximum possible distance must be reached before losing balance. During the test, you must move the object consecutively on each axis, without resting the other foot on the ground, until you travel the 3 strips. At this time, the test will end and the evaluator will measure the distance traveled. The subject will be urged to repeat the test again, up to a total of 3 times. Next, the same procedure will be performed with the contralateral member.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain